CLINICAL TRIAL: NCT01001429
Title: Comparison of Dexmedetomidine vs. Propofol in Vitreoretinal Surgery Under Sub-Tenon's Block
Brief Title: Dexmedetomidine Versus Propofol in Vitreoretinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0120090202
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-04

CONDITIONS: Retinal Detachment
Keywords: sedation for vitreoretinal surgery
MeSH Terms: conditions — Retinal Detachment | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): propofol 1mg/kg as a bolus intravenously followed by an infusion of 25-100 ug/kg/min
  Interventions: Drug: propofol
- dexmedetomidine infusion (Experimental): Subject will receive a bolus of0.5ug/kg intravenously over a period of 10-15 minutes, followed by an infusion of 0.2-0.7ug/kg/hr of drug.
  Interventions: Drug: Dexmedetomidine infusion

INTERVENTIONS:
Drug: Dexmedetomidine infusion — bolus of 0.5ug/kg intravenously over a period of 10-15 minutes, followed by an infusion of 0.2-0.7ug/kg/hr of drug
  Other Names: Precedex infusion
  Arms: dexmedetomidine infusion
Drug: propofol — propofol 1mg/kg intravenously as a bolus followed by 25-100ug/kg/min
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
The investigators would like to determine if using Dexmedetomidine alone or in a reduced dose can prevent or reduce the incidence of adverse effects, while providing adequate sedation, and respiratory stability as compared to propofol.

DETAILED DESCRIPTION:
Alpha2 adrenergic receptor agonist have been used increasingly as a new armamentarium to provide sedative/hypnotic, analgesic, anxiolytic and sympatholytic effects in the perioperative settings. Dexmedetomidine, a selective and specific alpha2- adrenoceptor agonist has unique properties that makes it an almost ideal sedative drug for monitored anesthesia care in procedures under local or regional block. Unlike other drugs use for sedation, dexmedetomidine induces sedation that is similar to natural sleep (readily arousable) without causing respiratory depression. It attenuates the stress-induced sympathoadrenal response seen with laryngoscopy and intubation. It has anesthetic and opioid sparing effects, hence it may be a useful adjunct to general anesthesia and monitored anesthesia care in patients susceptible to narcotic induced respiratory depression. Another unique property of dexmedetomidine is that its sedative effect is reversible with Atipamezole. A previous study wherein dexmedetomidine has been used in procedures under local and regional block had shown that it provides effective sedation and better operating condition without significant respiratory depression. As a supplement to general anesthesia, it has been shown to provide stable hemodynamics. However, it is associated with some adverse events such as hypertension, hypotension and bradycardia, these commonly occur during bolus administration of the recommended dose of 1ug/kg. Post-operatively it can cause nausea and vomiting. Vitreoretinal surgery requires either an injection of local anesthetic within the muscle cone (retrobulbar block),or into the periorbital space (peribulbar block). This can be done individually or in combination. This surgery can also be done under a safer technique of retrobulbar block that is given using a sub-tenon's approach through a snip peritomy; a blunt cannula can be used with this technique mitigating the complications of retrobulbar hemorrhage or inadvertent injection into the optic nerve sheath or perforation of the globe using a sharp needle. The anesthetic goal is to provide an immobile and uncongested operative field. Hemodynamic stability of the patient is also important since some patients that require this procedure are elderly with co-morbid conditions such as hypertension, diabetes mellitus and Coronary Artery Disease (CAD). In our study we would like to investigate if Dexmedetomidine alone and in a reduced dose can prevent or reduce the incidence of adverse effects, provide hemodynamic and respiratory stability, provide adequate sedation with patient and surgeon satisfaction and compare it with Propofol.

Objectives:

Primary:

1. Adequate sedation
2. Hemodynamic and respiratory stability intraoperatively

Secondary:

1. surgeon satisfaction
2. Time to achieved " street fitness " status
3. subject satisfaction
4. Hemodynamic stability in PACU

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists rating of I-III
* good renal and liver function

Exclusion Criteria:

* renal and hepatic insufficiency
* uncontrolled diabetes
* uncontrolled hypertension
* severe cardiac disease Class III or IV
* heart blocks
* chronic use of sedatives, narcotics, alcohol or illicit drugs
* allergy to either propofol or dexmedetomidine
* pregnancy or inability to tolerate technique of the study drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Patel, MD, Principal Investigator — Rutgers /NJMS
Locations (2):
- United States (2):
  - UMDNJ-University Hospital, Newark, New Jersey
  - University Hospital, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited the morning of surgery in the Same Day Surgery Suite
Pre-assignment Details: One subject withdrew consent prior to group assignment. One subject surgery was cancelled
Period: Overall Study
Arm/Group | Propofol | Dexmedetomidine Infusion
Started | 39 | 38
Completed | 39 | 37
Not Completed | 0 | 1
Not completed — surgery cancelled | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Dexmedetomidine Infusion | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 40 [40 to 60] | 52 [42.8 to 61.2] | 46 [40 to 61.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 28 | 25 | 53
total participants [Number; unit: participants] | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Adequate Sedation Via Bispectral Index Score (BIS)and University of Michigan Sedation Scale (UMSS)
Description: Bispectral Index Score measurement uses processed electroencephalogram signals to measure sedation depth of a scale from 0-100 (0=coma; 40-60=general anesthesia;60-90 sedated;100=awake) University of Michigan Sedation Scale (1-4) is an observational scale that quantifies sedation.1=normal response to verbal stimuli, 2=conscious sedation, responsive to tactile stimuli, 3= deeply sedated responsive to repeated or painful stimuli, 4=general anesthesia: not arousable.
Time Frame: Intraoperative up to 120 min
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Groups:
- BIS Scores in Propofol Infusion Group: propofol 1mg/kg as a bolus intravenously followed by an infusion of 25-100 ug/kg/min
  propofol: propofol 1mg/kg intravenously as a bolus followed by 25-100ug/kg/min
- BIS Scores in Dexmedetomidine Infusion Group: Subject will receive a bolus of 0.5ug/kg intravenously over a period of 10-15 minutes, followed by an infusion of 0.2-0.7ug/kg/hr of drug.
  Dexmedetomidine infusion: bolus of 0.5ug/kg intravenously over a period of 10-15 minutes, followed by an infusion of 0.2-0.7ug/kg/hr of drug
- UMSS Scores in Propofol Infusion Group: Propofol medication administered as described in BIS group/Propofol group
- UMSS in Dexmedetomidine Infusion Group: subject received medication as described in BIS/dexmedetomidine
Arm/Group | BIS Scores in Propofol Infusion Group | BIS Scores in Dexmedetomidine Infusion Group | UMSS Scores in Propofol Infusion Group | UMSS in Dexmedetomidine Infusion Group
Number analyzed (Participants) | 39 | 37 | 39 | 37
units on a scale | 84.8 [77.5 to 92.1] | 88 [78 to 94] | .90 [.47 to 1.33] | .94 [.43 to 1.45]
Statistical Analysis 1: Comparison: BIS Scores in Propofol Infusion Group vs BIS Scores in Dexmedetomidine Infusion Group; Test type: Superiority or Other; p = 0.04, Regression, Logistic
Statistical Analysis 2: Comparison: UMSS Scores in Propofol Infusion Group vs UMSS in Dexmedetomidine Infusion Group; UMSS scores with subjects propofol vs. Dexmetomidine group; Test type: Superiority or Other; p = 0.68, Regression, Linear

2. Secondary Outcome: Time to Achieve "Street Fitness"
Description: Subjects will be kept in the Post Anesthesia Care Unit (PACU) for a period of 2 hours. However it will be documented as to when, in the opinion of the PACU staff, the subject has met the criteria for discharge.
Time Frame: for 2 hours post-operatively in Post Anesthesia Care unit
Population: Subjects meet criteria for discharge based upon the assessment from a professional independent of the study
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Propofol | Dexmedetomidine Infusion
Number analyzed (Participants) | 39 | 37
minutes | 81 [54 to 108] | 85 [49.8 to 120]

3. Primary Outcome: Intraoperative Hemodynamic Stability
Description: systolic and diastolic blood pressure was recorded at 5 minute intervals up to 120 min and were averaged per study arm
Time Frame: Intraoperative up to 120 min
Measure: Mean (Inter-Quartile Range); unit: mm/Hg
Groups:
- Propofol Group -Mean Systolic Blood Pressure: propofol 1mg/kg as a bolus intravenously followed by an infusion of 25-100 ug/kg/min
  propofol: propofol 1mg/kg intravenously as a bolus followed by 25-100ug/kg/min
- Dexmedetomidine Group-mean Systolic Blood Pressure: Subject will receive a bolus of0.5ug/kg intravenously over a period of 10-15 minutes, followed by an infusion of 0.2-0.7ug/kg/hr of drug.
  Dexmedetomidine infusion: bolus of 0.5ug/kg intravenously over a period of 10-15 minutes, followed by an infusion of 0.2-0.7ug/kg/hr of drug
- Propofol Group- Mean Diastolic Blood Pressure: propofol administered as described- blood pressure recorded at 5 min intervals during surgery
- Dexmedetomidine Group- Mean Diastolic Blood Pressure: dexmedetomidine as already described and blood pressure monitored 5 min intervals,
Arm/Group | Propofol Group -Mean Systolic Blood Pressure | Dexmedetomidine Group-mean Systolic Blood Pressure | Propofol Group- Mean Diastolic Blood Pressure | Dexmedetomidine Group- Mean Diastolic Blood Pressure
Number analyzed (Participants) | 39 | 37 | 39 | 37
mm/Hg | 124.9 [108.7 to 141.1] | 114.6 [100.1 to 129.1] | 73.6 [61.1 to 86.1] | 66.2 [55.4 to 77.0]

4. Primary Outcome: Intraoperative Respiratory Stability
Description: respiratory rate data were recorded at 5 minutes intervals throughout the surgical procedure up to 120 mins for both groups and averaged per study arm
Time Frame: Intraoperative up to 120 min
Measure: Mean (Full Range); unit: breaths per minute
Groups:
- Propofol Group: subjects randomized to propofol group had their respiratory rate recorded at 5 minute intervals during the operative procedure.
- Dexmedetomidine Group: subjects randomized to dexmedetomidine group had their respiratory rate recorded at 5 minute intervals during the operative procedure
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 39 | 37
breaths per minute | 17 [12 to 22] | 12 [8 to 16]

5. Primary Outcome: Intraoperative Heart Rate Stability
Description: Heart rate recorded at 5 minute intervals during surgery up to 120 min and averaged per study arm
Time Frame: Intraoperative up to 120 min
Measure: Mean (Full Range); unit: beats per minute
Groups:
- Propofol Group: Heart rate recorded at 5 minute intervals during procedure for subjects randomized to propofol
- Dexmedetomidine: Heart rate recorded at 5 minute interval for subjects randomized to dexmedetomidine
Arm/Group | Propofol Group | Dexmedetomidine
Number analyzed (Participants) | 39 | 37
beats per minute | 71 [58 to 84] | 64 [49 to 80]

6. Secondary Outcome: Surgeon Satisfaction for Adequate Sedation
Description: 1=very poor, 2=poor,3=fair, 4=good, 5=excellent
Time Frame: at 10 minutes into the procedure
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Propofol Group: surgeon satisfaction at 10 minutes in to the procedure for subjects randomized to propofol
- Dexmedetomidine Group: surgeon satisfaction at 10 minutes into the procedure
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 39 | 37
units on a scale | 4.62 [3 to 5] | 4.97 [3 to 5]

7. Secondary Outcome: Surgeon Satisfaction for Adequate Sedation at Completion of Procedure
Description: surgeon satisfaction graded on numerical scale 1=very poor. 2=poor, 3=fair 4=good, 5=excellent
Time Frame: immediately following the completion of the procedure up to one hour
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Propofol Group: patients receiving comparison drug propofol
- Dexmedetomidine Group: patients receiving study drug dexmedetomidine
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 39 | 37
units on a scale | 4.77 [3 to 5] | 4.89 [3 to 5]

8. Secondary Outcome: Patient Satisfaction
Description: 1=very poor, 2=poor, 3=fair, 4=very good, 5=excellent
Time Frame: measured prior to discharge up to 2 hours
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Propofol: patient satisfaction prior to discharge on a 5 point scale1=very poor, 2=poor, 3=fair, 4= good , 5=excellent
- Dexmedetomidine Group: patient satisfaction
  1=very poor, 2=poor, 3=fair, 4= good, 5=excellent
Arm/Group | Propofol | Dexmedetomidine Group
Number analyzed (Participants) | 39 | 37
units on a scale | 4.61 [3 to 5] | 4.43 [3 to 5]

9. Secondary Outcome: Post Operative Hemodynamic Stability
Description: blood pressure documented at 30 minute intervals in PACU up to 120 min
Time Frame: 2 hours in PACU
Measure: Mean (Inter-Quartile Range); unit: mmHg
Groups:
- Propofol Group: systolic blood pressure at 30 min intervals in PACU
- Dexmedetomidine Group: systolic blood pressure measured at 3 0 min. intervals in PACU
- Propofol: diastolic blood pressure recorded every 30 min in PACU
- Dexmedetomidine: diastolic pressure measured every 30 min in PACU
Arm/Group | Propofol Group | Dexmedetomidine Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 39 | 37 | 39 | 37
mmHg | 124.9 [108.7 to 141.1] | 114.6 [100.1 to 129.1] | 73.6 [61.1 to 86.1] | 66.2 [55.4 to 77]

10. Secondary Outcome: Hemodynamic Stability Post Operatively in PACU
Description: heart rate recorded at 30 min intervals in PACU up to 120 min
Time Frame: PACU to 2 hours post op
Measure: Mean (Inter-Quartile Range); unit: beats per minute
Groups:
- Propofol Group: heart rate recorded in 30 min intervals in PACU ( 2 hours)
- Dexmedetomidine: heart rate recorded at at 30 min intervals while in PACU (2 hours)
Arm/Group | Propofol Group | Dexmedetomidine
Number analyzed (Participants) | 39 | 37
beats per minute | 74.1 [72 to 77] | 72 [71 to 73]

ADVERSE EVENTS:
Time Frame: Heart rate, blood pressure, pulse oximetry are collected for all patients undergoing sedation or anesthesia for the entire time they are in the operating room which was between 1-2 hrs. Additionally heart rate, blood pressure, pulse oximetry were monitored for 2 hours in the Post Anesthesia Care Unit where patients are placed immediately following the procedure.
Description: Change in ECG, T wave inversion was noted on the cardiac monitor in the operating room, no intervention was required and the surgery continued without incident. A cardiology consult was called and the subject was admitted for observation. A myocardial perfusion test demonstrated a fixed deficit in the left ventricle, the Ejection fraction was 55% and serial Troponin levels were<0.2, well below threshold for evidence of myocardial injury
Arm/Group | Propofol | Dexmedetomidine Infusion
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/37
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=39) | Dexmedetomidine Infusion (N=37)
T wave inversion on EKG (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Termination of study due to difficulty recruiting subjects who fit the study criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes